CLINICAL TRIAL: NCT06224374
Title: Validity and Reliability of the Newly Developed Balance Assessment System in Healthy Young Adults
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Elcin Akyurek, Principal Investigator, Istanbul University - Cerrahpasa
Other Study IDs: AkyurekE3
Record Dates: First submitted 2024-01-16; First posted 2024-01-25 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Healthy; Assessment, Self
Keywords: young adult; healthy; balance; validity; assessment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Validity and Reliability: Participants will be evaluated with the "Postural Stability Test", "Limits of Stability Test", "Sensory Integration Test" and "Bilateral Comparison Test" within the AlBalance and Biodex Balance Evaluation System. To calculate the test-retest reliability and validity of the devices, these measurements will be made by the same evaluator in two sessions, 7 days apart. To eliminate the learning effect, participants who try AlBalance first in the first session will be the first to try Biodex in the second session (reverse test order will be used). Participants who complete all evaluations with the first device will rest for 5 minutes and move on to the other device. Then, parallel clinical tests will be applied to the participants, "Functional Reaching Test" and "One Leg Standing Test". The relationship of outcome measurements between devices and measurements of each test will be evaluated with statistical methods.

SUMMARY:
The goal of this observational study is to to evaluate the validity and reliability of the "Postural Stability Test", "Stability Limits Test", "Sensory Integration Test" and "One-Leg Standing Test" tests of the newly developed patented balance assessment system in healthy young adults. The main questions it aims to answer are:

* Are the "Postural Stability Test", "Stability Limits Test", "Sensory Integration Test" and "One-Leg Standing Test" tests in the newly developed balance assessment system a valid method for healthy young adults?
* Are the "Postural Stability Test", "Stability Limits Test", "Sensory Integration Test" and "One-Leg Standing Test" tests in the newly developed balance assessment system a reliable method for healthy young adults?

Participants will be evaluated with the "Postural Stability Test", "Limits of Stability Test", "Sensory Integration Test" and "Bilateral Comparison Test" within the AlBalance Balance Evaluation System and Biodex Balance Evaluation System. Participants will be asked to sit in a chair and rest for 5 minutes before starting the tests. To calculate the test-retest reliability and validity of the devices, these measurements will be made by the same evaluator in two sessions, 7 days apart. To eliminate the learning effect, participants who try AlBalance first in the first session will try Biodex first in the second session (reverse test order will be used). Participants who complete all evaluations with the first device will rest for 5 minutes and move on to the other device. Then, parallel clinical tests will be applied to the participants, "Functional Reaching Test" and "One Leg Standing Test".

DETAILED DESCRIPTION:
Balance refers to the ability to maintain the center of gravity within the base of support, regardless of age, and is the foundation of movement. Postural stability is defined as the ability to control the body's center of mass on the base of support and maintain an upright posture. Postural stability is a complex skill that relies on the interaction of multiple dynamic sensorimotor and cognitive systems under static and dynamic conditions. Postural stability and balance are two of the most important factors that determine a person's ability to make and maintain movements Conducting balance and postural stability research is of great importance for both diagnosis and treatment purposes. Commonly used tests such as the Berg Balance Test and Functional Reaching Test can detect changes in balance and postural stability, but the accuracy of the tests is limited as they are highly dependent on the tester's abilities and familiarity with the scale. Therefore, in addition to clinical evaluations, various commercial testing devices are also used to provide needed information about balance and postural stability. Our study aims to evaluate the validity and reliability of the "Postural Stability Test", "Limits of Stability Test", "Sensory Integration Test" and "Bilateral Comparison Test" tests of the newly developed patented balance assessment system in healthy young adults.

With this study, the reliability of a new and local balance assessment system will be tested in healthy young adults. We think that this study will provide preliminary information about the use of a new and local device for professionals working in the field of postural stability and balance assessment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-25
* Body mass index is below 24
* They should be able to understand and follow instructions
* Volunteering to participate in the study

Exclusion Criteria:

* Presence of neuromuscular, rheumatic disease or vestibular problems that may affect balance
* Having a visual impairment that affects vision
* Any other exercise or physical activity that may affect trunk muscle strength or balance
* Having a recent history of orthopedic injury or surgery in the lower extremity
* Having experienced any acute situation that could affect postural stability and balance between the two tests (within 7 days)

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young adult between the ages of 18-25 who meet the inclusion criteria will be included in our study.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Postural Stability Test | Change from baseline to 7 day
  Stability indices represent fluctuations around the zero point established before testing when the platform is stable. With the "Postural Stability Test", the anteroposterior, right-left, and general stability indexes of the cases will be recorded. During the test, participants will be asked to stand on the force platform with their feet in a comfortable position, arms at their sides, and palms facing toward the thighs. All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. The participant will be asked to stand still looking at the screen in front of him for 30 seconds. In both devices, there will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's postural stability will be assessed with postural stability test.
Limits of Stability | Change from baseline to 7 day
  In this test, the participant stands on force plates and deliberately shifts his or her body weight in the direction indicated on the screen without lifting his or her feet off the ground. This protocol measures various movement characteristics in 8 different directions: front, forward/right, right, back/right, back, back/left, left, and forward/left. During the test, participants will be asked to stand on the force platform with their feet in a comfortable position, arms at their sides, and palms facing toward the thighs. Direction control (%) and test times (sec) in all directions of the participants, who will move in 8 different directions sequentially, will be recorded. In both devices, there will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's limits of stability will be assessed with limits of stability test.
Sensory Integration Test | Change from baseline to 7 day
  The test decides which of the visual, vestibular, and proprioceptive information is used to provide orientation to maintain balance in different situations. During the test, visual and proprioceptive stimuli are disrupted and the ability to maintain the center of gravity is evaluated. The test consists of 4 different situations that gradually become more difficult: Situation 1: Eyes open; firm surface Situation 2: Eyes closed; firm surface Situation 3: Eyes open; foam surface Situation 4: Eyes closed; foam surface All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. The participant will be asked to stand still looking at the screen in front of him for 30 seconds. In both devices, there will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's sensory integration will be assessed with Sensory Integration Test.
Bilateral Comparison Test | Change from baseline to 7 day
  Bilateral Comparison test demonstrates postural stability by measuring the individual's ability to stand on one leg with eyes open and closed. On the balance platform, the individual stands on one leg with his hands at hip level. The test is repeated for the right foot and left foot. For both feet, 3 trials with eyes open and 3 trials with eyes closed are made. Each trial lasts 30 seconds. What is required from the individual is to remain stable on one leg as much as possible without losing balance. All measurements will be made with bare feet, and without shoes, and foot position will be recorded using coordinates on the platform's grid to ensure consistency in testing. In both devices, there will be a 1-minute rest break between measurements and they will be performed 3 times. The participant's bilateral comparison will be assessed with Bilateral Comparison Test.
Multimodal Functional Reach Test | Change from baseline to 7 day
  Multimodal functional reaching test is performed in three different positions: front, back, and side.
  In the functional forward reach test, the patient stands with the arm flexed at 90° and the fist closed, not touching but close to the wall. Three attempts are made and the average of these attempts is taken.
  In the functional back reach test, the patient stands with the arm flexed at 90° and the fist closed, not touching but close to the wall. Three attempts are made and the average of these attempts is taken.
  In the functional lateral reach test, the patient stands with his back to the wall, without touching the wall, keeping his arm in 90° abduction and his fist closed. Three attempts are made and the average of these attempts is taken. Multimodal Functional Reach Test will performed as parallel clinical tests and the participant's Multimodal Functional Reach will be assessed with Multimodal Functional Reach Test.
One Leg Stance Test | Change from baseline to 7 day
  The one-leg stance test demonstrates postural stability by measuring the individual's ability to stand on one leg with eyes open and closed. The individual stands on one leg with his hands at hip level. The test is repeated for the right foot and left foot. For both feet, 3 trials with eyes open and 3 trials with eyes closed are made. Each trial lasts 30 seconds. What is required from the individual is to remain stable on one leg as much as possible without losing balance. One Leg Stance Test will performed as parallel clinical tests and the participant's One Leg Stance will be assessed with One Leg Stance Test.

CONTACTS AND LOCATIONS:
Overall Officials: Asena Yekdaneh, Principal Investigator — Fenerbahçe University; İrem Kurt Ulusoy, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Elçin Akyürek, Principal Investigator — Istanbul University-Cerrahpasa, Institute of Postgraduate Education; Nilay Arman, Study Chair — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Ayşe Zengin Alpözgen, Principal Investigator — Istanbul University-Cerrahpaşa Faculty of Health Sciences; Bülent Bayraktar, Principal Investigator — Istanbul Faculty of Medicine, Department of Internal Medical Sciences, Department of Sports Medicine